CLINICAL TRIAL: NCT01243398
Title: Phase III Randomized, Double-Blind, Placebo-Controlled Trial of Gefitinib (Iressa®) Versus Placebo in Esophageal Cancer Progressing After Chemotherapy
Brief Title: Gefitinib in Treating Patients With Esophageal Cancer That is Progressing After Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDR0000689080; OXFORD-COG; UO-COG; EUDRACT-2007-005391-13; ISRCTN-29580179; AZ-D7913L00059; EU-21085
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Esophageal Cancer
Keywords: adenocarcinoma of the gastroesophageal junction; adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; recurrent esophageal cancer; stage IA esophageal cancer; stage IB esophageal cancer; stage IIA esophageal cancer; stage IIB esophageal cancer; stage IIIA esophageal cancer; stage IIIB esophageal cancer; stage IIIC esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gefitinib 500mg once daily (Experimental): Gefitinib 500mg once daily
  Interventions: Procedure: quality-of-life assessment
- Placebo (Placebo Comparator): Gefitinib 500mg once daily
  Interventions: Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether gefitinib is more effective than a placebo in treating esophageal cancer.

PURPOSE: This randomized phase III trial is studying gefitinib to see how well it works compared with a placebo in treating patients with esophageal cancer that is progressing after chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess whether gefitinib vs placebo will improve overall survival of patients with esophageal or gastroesophageal junction cancer.

Secondary

* To assess the toxicity of gefitinib monotherapy in these patients.
* To assess whether gefitinib vs placebo will have a significant positive or negative impact upon quality of life of these patients.
* To assess the impact gefitinib vs placebo will have on progression-free survival of these patients.

OUTLINE: This is a multicenter study.

* Arm A: Patients receive oral gefitinib once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.
* Arm B: Patients receive oral placebo once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

Blood samples are collected for genetic and translational studies. Patient's quality of life is assessed at baseline and periodically during the study with completion of EORTC Quality of Life Questionnaire (QLQ-C30) version 3.0.

After completion of study treatment, patients are followed up every 8 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed esophageal cancer or gastroesophageal junction tumor including the following subtypes:

  * Adenocarcinoma
  * Squamous cell cancer
  * Poorly differentiated epithelial malignancy
  * Gastroesophageal junction with Siewert type I or II tumors
* Failure after no more than 2 prior chemotherapy regimens and 1 chemoradiation course
* Measurable or evaluable disease by CT scan
* Patients with brain metastases must be stable and have received cranial irradiation prior to entry

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Serum bilirubin ≤ 3 times the upper limit of normal (ULN)
* AST/ALT ≤ 2.5 times ULN (≤ 5 x in presence of liver metastases)
* Able to take oral tablets (whole or dispersed)
* No evidence of clinically active interstitial lung disease (patients with chronic, stable, radiographic changes who are asymptomatic allowed)
* No known severe hypersensitivity to gefitinib or any of the excipients of this product
* No prior other malignancy likely to confound results or interfere with gefitinib therapy
* No medical condition considered to interfere with the safe participation in the trial
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No chemotherapy (including oral) within the past 6 weeks
* No radiotherapy to site of measurable or evaluable disease within the past 4 weeks
* No other concurrent cytotoxic chemotherapy, immunotherapy, hormonal therapy (excluding contraceptives and replacement steroids) or experimental medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2009-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Overall survival | 4, 8, 12, 16 weeks then every 8 weeks

SECONDARY OUTCOMES:
Toxicity and safety | 4, 8, 12, 16 weeks then every 8 weeks
Quality of life | 4, 8 and 12 weeks
Progression-free survival | 4, 8, 12, 16 weeks then every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Ferry, MD, Principal Investigator — New Cross Hospital
Locations (1):
- New Cross Hospital, Wolverhampton, England, United Kingdom